CLINICAL TRIAL: NCT00681447
Title: A Randomized, Prospective, Double-Blind Controlled Evaluation of the Effectiveness of Lumbar Interlaminar Epidural Injections in Lumbar Disc Herniation, and Discogenic Pain
Brief Title: Treatment of Chronic Low Back and Lower Extremity Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pain Management Center of Paducah (Other)
Responsible Party: Principal Investigator, Laxmaiah Manchikanti, MD, Medical Director, Pain Management Center of Paducah
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: protocol 15
Record Dates: First submitted 2008-03-14; First posted 2008-05-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Low Back Pain
Keywords: lumbar disc herniation; discogenic pain; lumbar interlaminar epidural; injections
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I (Other): Lumbar interlaminar epidural injection with local anesthetic only
  Interventions: Procedure: Lumbar Interlaminar Epidural; Procedure: Lumbar Interlaminar Epidural injection
- Group II (Other): Lumbar Interlaminar Epidural Injection with local anesthetic wiht 6 mg of non-particulate Celestone
  Interventions: Procedure: Lumbar Interlaminar Epidural; Procedure: Lumbar Interlaminar Epidural injection

INTERVENTIONS:
Procedure: Lumbar Interlaminar Epidural — 1. Lumbar interlaminar epidural injections under fluoroscopy
  2. Epidural tray and needle
  3. Drugs:
  0.5% Xylocaine and non-particulate Celestone
Procedure: Lumbar Interlaminar Epidural injection — 1. Lumbar interlaminar epidural injections under fluoroscopy
  2. Epidural tray and needle
  3. Drugs:
  0.5% Xylocaine and non-particulate Celestone

SUMMARY:
1. To demonstrate clinically significant improvements in patients undergoing lumbar interlaminar epidurals. Improvement will be assessed in relation to the clinical outcome measures of pain and function.
2. To evaluate and compare the adverse event profile in all patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of at least 18 years of age
* Subjects with a history of chronic, function-limiting chronic low back pain of at least 6 months in duration
* Subjects who are able to give voluntary, written informed consent to participate in this investigation
* Subjects who, in the opinion of the PI, are able to understand this investigation, co-operate with the investigational procedures, and are willing to return to the center for all the required post-operative follow-ups
* Subjects have not had recent surgical procedures within the last 3 months.

Exclusion Criteria:

* Cauda Equina symptoms and/or compressive radiculopathy
* Narcotic use of no greater than hydrocodone 100 mg/day, methadone of 60 mg, or morphine 180 mg, or dose equivalent
* Uncontrolled major depression or uncontrolled psychiatric disorders
* Uncontrolled or acute medical illnesses including coagulopathy, renal insufficiency, chronic liver dysfunction, progressive neurological deficit, urinary sphincter dysfunction, infection, increased intracranial pressure, pseudotumor cerebri, intracranial tumors, unstable angina, and severe chronic obstructive pulmonary disease.
* Chronic severe conditions that could interfere with the interpretations of the outcome assessments for pain and bodily function
* Women who are pregnant or lactating
* Subjects who have participated in a clinical study with an investigational product within 30 days of enrollment
* Patients with multiple complaints involving concomitant hip osteoarthritis, due to the overlap of pain complaints
* Inability to achieve appropriate positioning and inability to understand informed consent and protocol
* History of adverse reaction to local anesthetic or anti-inflammatory drugs and history of gastrointestinal bleeding or ulcers
* Previous surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-02; Primary Completion 2010-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate clinically significant improvement or lack thereof with the lumbar interlaminar epidural patients with or without steroids. | Patients will return for follow-up visits at 3, 6, 12, 18, and 24 months post-treatment. The recruitment period is estimated as 24 months with an anticipated study duration of 48 months.

SECONDARY OUTCOMES:
To evaluate differences in outcomes in patients receiving steroids compared to those patients randomized to the local anesthetic group who did not receive steroids. | Patients will return for follow-up visits at 3, 6, 12, 18, and 24 months post-treatment. The recruitment period is estimated as 24 months with an anticipated study duration of 48 months.
To evaluate and compare the adverse event profile in all patients. | Patients will return for follow-up visits at 3, 6, 12, 18, and 24 months post-treatment. The recruitment period is estimated as 24 months with an anticipated study duration of 48 months.

CONTACTS AND LOCATIONS:
Overall Officials: Laxmaiah Manchikanti, MD, Principal Investigator — Ambulatory Surgery Center, Paducah
Locations (1):
- Ambulatory Surgery Center, Paducah, Kentucky, United States

REFERENCES:
- [Derived] Manchikanti L, Cash KA, McManus CD, Damron KS, Pampati V, Falco FJ. A randomized, double-blind controlled trial of lumbar interlaminar epidural injections in central spinal stenosis: 2-year follow-up. Pain Physician. 2015 Jan-Feb;18(1):79-92. PMID 25675062
- [Derived] Manchikanti L, Singh V, Cash KA, Pampati V, Falco FJ. A randomized, double-blind, active-control trial of the effectiveness of lumbar interlaminar epidural injections in disc herniation. Pain Physician. 2014 Jan-Feb;17(1):E61-74. PMID 24452658
- [Derived] Manchikanti L, Cash KA, McManus CD, Pampati V, Benyamin RM. A randomized, double-blind, active-controlled trial of fluoroscopic lumbar interlaminar epidural injections in chronic axial or discogenic low back pain: results of 2-year follow-up. Pain Physician. 2013 Sep-Oct;16(5):E491-504. PMID 24077199
- [Derived] Manchikanti L, Cash KA, McManus CD, Damron KS, Pampati V, Falco FJ. Lumbar interlaminar epidural injections in central spinal stenosis: preliminary results of a randomized, double-blind, active control trial. Pain Physician. 2012 Jan-Feb;15(1):51-63. PMID 22270738
- [Derived] Manchikanti L, Cash KA, McManus CD, Pampati V, Benyamin RM. Preliminary results of a randomized, double-blind, controlled trial of fluoroscopic lumbar interlaminar epidural injections in managing chronic lumbar discogenic pain without disc herniation or radiculitis. Pain Physician. 2010 Jul-Aug;13(4):E279-92. PMID 20648214
- [Derived] Manchikanti L, Singh V, Falco FJ, Cash KA, Pampati V. Evaluation of the effectiveness of lumbar interlaminar epidural injections in managing chronic pain of lumbar disc herniation or radiculitis: a randomized, double-blind, controlled trial. Pain Physician. 2010 Jul-Aug;13(4):343-55. PMID 20648203